CLINICAL TRIAL: NCT00689832
Title: Comparative, Multicentre, Randomised, Double-blind Study to Assess the Efficacy of Tacrolimus 0.03% Ointment Versus Fluticasone 0.005% Ointment in Children Aged 2 Years or Over Suffering From Moderate to Severe Atopic Dermatitis.
Brief Title: Protopic Ointment in Children Atopic Eczema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-506-06-FR-05; EUDRACT #:2004-002478-47
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Dermatologic Agents; Topical Drug Administration; Tacrolimus; Calcineurin; Corticosteroid; Fluticasone propionate; Child
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Tacrolimus 0.03%
- B (Active Comparator)
  Interventions: Drug: Fluticasone 0.005%

INTERVENTIONS:
Drug: Tacrolimus 0.03% — ointment
  Other Names: Protopic® 0.03%
  Arms: A
Drug: Fluticasone 0.005% — ointment
  Other Names: Flixovate® 0.005%
  Arms: B

SUMMARY:
Children with atopic eczema and a poor response to topical corticosteroid applied either Protopic or Fluticasone ointment twice a day for 3 weeks. They could continue during 3 more weeks once a day if needed.

DETAILED DESCRIPTION:
Treatments were to be applied twice daily until clearance, for a maximum of 3 weeks and then, in case of uncleared residual lesions, once daily for up to 3 further weeks. In the event of a flare-up the treatment was to be resumed twice a day until the end of the study.

Statistical methods: An interim analysis was performed on 30% of the planned total sample size, i.e. 140 included patients who had completed the study, to reassess the assumptions made during the planning phase.

ELIGIBILITY:
Inclusion Criteria:

* Children with moderate to severe atopic dermatitis (Rajka & Langeland score greater than or equal to 4.5) and who had responded insufficiently to conventional therapies
* Female patients of childbearing age: effective means of contraception throughout the period of the study and for four weeks following the end of the study
* Informed consent
* Therapeutic washout for atopic dermatitis treatments

Exclusion Criteria:

* Genetic epidermal barrier defect, such as Netherton's syndrome, or suffering from erythroderma
* Any female patients who were pregnant or breast-feeding
* Clinical infection due to the VZV virus (varicella, zona), HSV1-2 viruses (herpes), verruca vulgaris or molluscum contagiosum
* Superinfected eczema
* Known hypersensitivity to macrolides or to any other excipient in tacrolimus ointment
* Known hypersensitivity to one of the agents contained in the fluticasone 0.005% ointment preparation
* Ulcerated lesions, of whatever type
* Moderate to severe acne or rosacea
* Patients participating at the same time in another clinical study or who have participated in another clinical study within 28 days of the start of this study
* substance abuse (including that of drugs and alcohol) or mental disorder/psychological state which, in the investigator's opinion, might interfere with the patient's follow-up
* Known serologically proven HIV positivity

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 487 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting at the week 3 visit (day 21) with an improvement of at least 60% in their modified Eczema Area and Severity Index (mEASI) in comparison to day 1 | 3 weeks

SECONDARY OUTCOMES:
mEASI and EASI scores at each visit and percentage change with respect to day 1 | 1 week and 3 weeks
Global assessment of clinical response by the physician at each visit after day 1 | 1 week and 3 weeks
Global assessment of clinical response by the patient/parents at each visit after day 1 | 1 week and 3 weeks
All clinical signs, including sleep quality, severity of pruritus and body surface area affected at each visit | 1 week and 3 weeks
Compliance with the treatment assessed from the patient's diary | 1 week and 3 weeks
Patient's quality of life assessed at day 1 and day 21 | 3 weeks
Incidence of adverse events during the study | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Paris, France